CLINICAL TRIAL: NCT05493410
Title: EFFECTS OF INSPIRATORY MUSCLE TRAINING ON INSPIRATORY MUSCLE STRENGTH AND ENDURANCE AND FUNCTIONAL CAPACITY OF POST-COVID-19 PATIENTS
Brief Title: EFFECTS OF INSPIRATORY MUSCLE TRAINING IN POST-COVID-19 PATIENTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Vila Velha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 49725921.6.0000.5064
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Covid19
Keywords: covid19; inspiratory muscle training (IMT); maximum inspiratory pressure (MIP); dynamic inspiratory muscle strength index (S-Index); inspiratory muscle endurance; respiratory physicaltherapy; pulmonary rehabilitation
MeSH Terms: conditions — COVID-19 | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants were split into two experimental groups:
  CONTROL GROUP (CG): Pulmonary rehabilitation protocol comprising muscle strengthening and aerobic training; TREATMENT GROUP (TG): Pulmonary rehabilitation protocol comprising muscle strengthening, aerobic training, and inspiratory muscle training using the POWERbreathe Classic Medic® device.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding in the distribution of participants will be guaranteed, as it will be carried out by a different researcher from the one who will treat the patients. In addition, the researchers who will collect and analyze the data will be different and blind to the experimental groups and types of intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TREATMENT GROUP (TG) (Experimental): Pulmonary rehabilitation protocol consisting of muscle strengthening, aerobic training, and IMT using the POWERbreathe Classic Medic® device - será comparado with the CONTROL GROUP (CG), which will not undergo IMT.
  Interventions: Other: TREATMENT GROUP (TG)
- CONTROL GROUP (CG) (Active Comparator): Pulmonary rehabilitation protocol consisting of muscle strengthening and aerobic training.
  Interventions: Other: CONTROL GROUP (CG)

INTERVENTIONS:
Other: TREATMENT GROUP (TG) — In addition to muscle strengthening and aerobic exercise, patients from the TG will undergo IMT for six weeks, performing two sets of 30 repetitions daily using the device POWERbreathe classic medic® (POWERbreathe International Ltd., Southam, United Kingdom). MIP will be measured in all patients before the intervention as described earlier, and patients will exercise at 40% MIP in the first week and 60% MIP in the subsequent five weeks. The patients will be instructed to inhale using the diaphragm muscle, trying to expand the rib cage to avoid using accessory muscles A nose clip will be used to ensure patients breathe exclusively through the training device.
  Other Names: inspiratory muscle training using the POWERbreathe Classic Medic® device; muscle strengthening; aerobic training
  Arms: TREATMENT GROUP (TG)
Other: CONTROL GROUP (CG) — For six weeks the CG will perform muscle strengthening through a sit and stand up from a chair routine, abduction of upper and lower limbs, and rowing; three sets of 10 repetitions of each exercise will be performed. Elastic tubes will be used, with elasticity defined by color and indicating the greatest resistance the participant can endure with an effort between 4 and 8 on the OMNI-RES scale for perceived exertion.
  In addition, aerobic exercise will be performed, through walking on flat terrain for five minutes in the first week, 10 minutes in the second week, and 20 minutes in the subsequent week, with intensity between 40-60% of the reserve heart rate and respecting the patients' symptoms.
  Aerobic training intensity will be calculated by the modified BORG exertion scale maintaining a score between 6 and 7 - with the progression respecting the patients' symptoms - and by the reserve heart rate.
  Other Names: muscle strengthening; aerobic training
  Arms: CONTROL GROUP (CG)

SUMMARY:
COVID-19 is an infectious disease caused by the SARS-CoV-2 virus, which had its first case identified in December 2019 in Wuhan, China. The disease can cause death and collapse in health systems, in addition to increasingly prevalent sequelae. Among the persistent symptoms presented by patients in the post-COVID-19 phase, we highlight the respiratory ones. The diaphragm - the main muscle of respiration - can also undergo structural and functional changes resulting from SARS-CoV-2 infection. This finding is related to some respiratory sequelae of the disease, such as severe myopathy of the diaphragm with weakness and decreased endurance of the inspiratory muscles, dyspnea, fatigue, and failure in ventilatory weaning. Considering that COVID-19 can affect the respiratory muscles of afflicted individuals, it is reasonable to assume that inspiratory muscle training should improve inspiratory muscle weakness and endurance, and the functional capacity of individuals who had symptomatic COVID-19. Objective: To evaluate the effect of inspiratory muscle training on inspiratory muscle strength and endurance and on the functional capacity of individuals afflicted by COVID-19. Methods: This controlled and randomized clinical trial will be conducted according to the guidelines of the Vila Velha University Ethics Committee (CEP-UVV). The sample will consist of individuals with a positive diagnosis for SARS-CoV-2 infection assessed by means of the reverse transcriptase reaction followed by the polymerase chain reaction (RT-PCR) and who have already undergone the period of active infection. These individuals will be invited to participate in the study as soon as they are evaluated by the cardiopulmonary rehabilitation service. Those who meet all the inclusion criteria, agree to participate, and sign the free and informed consent form (FICF), will be randomly assigned to two groups, the control group (CG, n = 21) and the treatment group (TG, n = 21). The initial evaluation will consist of anamnesis, measurement of indirect blood pressure, heart rate, and peripheral oxygen saturation by portable pulse oximeter, analysis of maximum inspiratory pressure (MIP), dynamic inspiratory muscle strength index (S-Index), and endurance of the inspiratory muscles - which will be collected using a digital training device (PowerBreathe KH2), in addition to functional assessment through the 1-minute sit-to-stand test. The reassessment will take place six weeks after the start of the program and the same data will be collected at the participants' homes. Both groups will undergo the rehabilitation protocol, consisting of muscle strengthening and aerobic training, with individual assessment of exercise intensity. The treated group will undergo inspiratory muscle training through linear pressure load, using the POWERbreathe Classic Medic® device to perform two sets of 30 repetitions daily for six weeks. The same physical therapist will oversee the training sessions of all patients. Statistical analysis: Data normality will be tested using the Shapiro-Wilk test. To analyze the differences between groups, we will use the t-test for parametric data and the Wilcoxon test for non-parametric data. The level of significance will be set at 5% (p < 0.05). Data will be analyzed using the SPSS 8.0 software and the results expressed as mean ± standard deviation or median and interquartile range.

DETAILED DESCRIPTION:
This randomized controlled clinical trial will be carried out according to the ethical standards for research with human beings and shall be previously approved by the human research ethics committee (CEP-UVV); participants will have to sign the free and informed consent form (FICF).

The sample will consist of individuals with a positive diagnosis for SARS-CoV-2 infection assessed by means of the reverse transcriptase reaction followed by the polymerase chain reaction (RT-PCR) and who have already undergone the period of active infection. The active infection period comprises 14 days from the onset of symptoms for those who have not been hospitalized and 21 days for those who have been hospitalized. These individuals will be invited to participate in the research as soon as they are evaluated by the cardiopulmonary rehabilitation service. Those who meet all the inclusion criteria, agree to participate, and sign the FICF will be randomly assigned to two groups, the control group (CG) and the treatment group (TG). The block randomization scheme will be generated using the randomization.com website (http://www.randomization.com). The allocation of participants will be carried out by a different researcher from the one who will treat the patients, thus ensuring blinding. In addition, the researchers who will collect and analyze the data will be different and both blind to the experimental groups and types of intervention.

Regarding the sample size, as the study was designed to detect a mean difference of 20 cmH2O in MIP between groups, with a standard deviation of 15 (Newall; Stockley, 2005), a 95% confidence level, and a significance level of 0.05 (two-tailed α), we calculated that each group should contain 15 subjects. Considering the possibility of a sample loss of 20-25%, 42 individuals will be recruited (21 per group). (Newall, 2005).

The initial assessment will be carried out by the cardiopulmonary rehabilitation service at home, in which the following data will be collected: anamnesis; blood pressure (BP) measurement by digital sphygmomanometer (Omron® HEM 705CP, Tokyo, Japão); heart rate (HR) and peripheral oxygen saturation (SpO2) by the portable pulse oximeter G-Tech Oled Graph® (Beijing Choice Electronic Technology Co., Ltd., Beijing, China); MIP, dynamic inspiratory muscle strength (S-Index), and inspiratory muscle endurance analyses using the POWERbreathe K-series KH2® (POWERbreathe International Ltd., Warwickshire, United Kingdom); and functional assessment through the 1-minute sit-to-stand test (1-min STS).

The reassessment will take place six weeks after the start of the program and the same data will be collected at the participants' homes.

The primary outcome of the study to evaluate inspiratory muscles will be MIP, while S-Index, endurance, and functional capacity will be secondary outcomes.

EVALUATION PROCEDURES:

1-MINUTE SIT-TO-STAND TEST This test assesses the functional capacity of individuals with different types of diseases or dysfunctions. This standardized assessment is performed in an armless, 46-cm-high chair. The individual evaluated receives the verbal command to get up and sit down from the chair as many times as possible within a 1-minute interval. The main outcome of the test is how many times the individual sat and stood up; secondarily, vital and perceived exertion data are recorded before, during, and immediately after the test is performed.

MEASUREMENT OF BP, HR, AND SPO2 BP will be measured using a digital sphygmomanometer (Omron® HEM 705CP, Tokyo, Japan). The patient will remain seated for five minutes in a comfortable chair, with the back relaxed and supported on the backrest, legs uncrossed, left arm supported on the table, and free of clothes at arm height. The patient cannot drink alcohol, have smoked or exercised 30 minutes before the measurement, and the bladder must be empty. Three measurements will be taken with a 2-min interval between them; the first will be discarded and the BP value obtained by the average between the last two measurements.

HR and SpO2 will be measured using the portable pulse oximeter G-Tech Oled Graph® (Beijing Choice Electronic Technology Co., Ltd., Beijing, China). Pulse oximetry measures how much oxygen the blood is carrying. Through a small device called a pulse oximeter, the blood oxygen level can be measured without the need for an arterial blood puncture. To measure oxygen, beams of light produced by the device pass through the blood on the finger and are "read" to calculate the percentage of oxygen transport. This method also measures HR. The accuracy of the oximeter is 2% above or 2% below the saturation that can be obtained by an arterial blood gas test. To obtain a better reading, the patient will be instructed to keep the hand warm, relaxed, kept below the level of the heart, and not to use fake nails and/or nail polish.

MIP, S-INDEX, AND ENDURANCE ANALYSES To analyze MIP, S-index, and endurance, we will use an electronic device employed by health professionals for the assessment and training of the inspiratory muscles in patients with dyspnea (POWERbreathe K series KH2®, HaB International, Warwickshire, United Kingdom). (POWERbreathe, 2019).

MIP assessment:

Initially, the patients will be instructed and familiarized with the device and the maneuver that will be performed, in which they will inhale against a closed airway, with prior warming of the inspiratory muscles and learning of the technique. MIP will be measured with the patients in a seated position. They will be encouraged to slowly exhale all the air and, from the residual volume (RV), perform a maximum inspiration. A nose clip and a mouthpiece with a bacteriological and viral filter, which must be well attached to the patient's mouth, will be used. Three maneuvers with 1-min rest intervals will be performed and recorded. Values must vary by less than 20%, and the highest one will be selected.

The MIP result displayed in the software corresponds to the highest 1-second mean pressure achieved during the maneuver (measured at 50 Hz). This measure reflects the pressure developed by the respiratory muscles plus the elastic recoil pressure of the respiratory system in the residual volume and is an index of global respiratory output rather than a direct measure of the contractile properties of the inspiratory muscles. This result will be used to monitor the influence of IMT.

The MIP values predicted for the Brazilian population have been published by several authors, and the main equations validated for Brazilians are the ones by: Neder et al.; Costa et al.; Simões et al., and Pessoa et al. The present proposal will predict MIP values through the equation of Neder et al., in which:

* For men: MIP (cmH2O) = 155,3 - (0,80 x age)
* For women: MIP (cmH2O) = 110,4 - (0,49 x age)

S-Index assessment:

The S-Index is a measure of the dynamic strength of the inspiratory muscles and is derived from the result of the peak inspiratory flow registered by the device's sensors in each incursion, using a patented algorithm. Unlike the isometric measurement (MIP), in this assessment the individual will perform the inspiratory maneuver through a valve with free air passage. Inspiratory muscle strength is calculated across the entire range of inspired lung volume. The result of the strength index is classified based on the normal values predicted for the population studied. These values, which are recorded in cmH2O, are individually calculated by the software Breathelink® (POWERbreathe, Warwickshire, United Kingdom), using information from the patient's profile. As patient learning has been described regarding this parameter, ten maneuvers will be performed in sequence, without rest between attempts, and the best result will be considered. The technique for measuring dynamic strength is similar to that of MIP, in which the patient must be seated, with a nose clip occluding the air passage through the nostrils, and a mouthpiece with a bacteriological and viral filter tightly coupled to the mouth.

Inspiratory muscle endurance assessment:

The tool POWERbreath K series® (POWERbreathe International Ltd., Warwickshire, United Kingdom) enables the performance of endurance tests (Silva et al, 2016). Endurance is the ability to sustain a specific task over time. The training load will be predetermined manually and introduced gradually over the first five breaths, as this is a constant load test, at 60% of the MIP value obtained from each patient. The patient will be instructed to breathe as long as possible until no breath can be fully completed, that is, until respiratory fatigue occurs. In the absence of respiratory fatigue, the maximum evaluation limit will be seven minutes, when the test is successfully completed. The results of resistance training will be recorded in the software and include the following parameters: Peak Inspiratory Flow (l/s), Training Load (cmH2O), Average Power (Watts), Average Inspired Volume (l), and Energy (Joules).

INTERVENTION CARDIOPULMONARY REHABILITATION All groups will undergo the rehabilitation protocol, comprised of muscle strengthening and aerobic training. Muscle strengthening will be achieved through a sit and stand up from a chair routine, abduction of upper and lower limbs, and rowing; three sets of 10 repetitions of each exercise will be performed. Elastic tubes will be used, with elasticity defined by color and indicating the greatest resistance the participant can endure with an effort between 4 and 8 on the OMNI-RES scale for perceived exertion (Tiggemann et al., 2010; Lagally, Robertson, 2006; Ramos et al., 2014; Ribeiro, 2021). In addition, aerobic exercise will be performed, through walking on flat terrain for five minutes in the first week, 10 minutes in the second, and 20 minutes in subsequent weeks, with intensity between 40-60% of the reserve heart rate and respecting the patients' symptoms (Spilmanns et al, 2021; Barker-Davies, 2020; Ribeiro, 2021) 3.6.1.1 Aerobic exercise intensity calculation

Aerobic training intensity will be calculated by the modified BORG subjective exertion scale maintaining a score between 6 and 7 - with the progression respecting the patients' symptoms - and by the reserve heart rate:

Target intensity = ((HRmax - HRrest) * 0.4 a 0.6) + HRrest First, maximum HR is determined using the Karvonen formula (220 - age) (KARVONEN, 1957).

On the day of the first assessment, the resting HR will be determined after the participant has been at rest for five minutes in a sitting position, in an environment at 22 oC. By determining HRmax and HRrest, it will be possible to calculate the target range for each participant. For individuals using beta blockers, the modified BORG subjective exertion scale will be used, maintaining a score between 6 and 7. The intensity and progression will be based on the individual reports of the symptoms of all patients (Spilmanns et al, 2021; Barker-Davies, 2020; Ribeiro, 2021).

3.6.2 INSPIRATORY MUSCLE TRAINING Patients from the TG will undergo IMT for six weeks, performing two sets of 30 repetitions daily using the device POWERbreathe classic medic® (POWERbreathe International Ltd., Southam, United Kingdom). MIP will be measured in all patients before the intervention as described earlier, and pa-tients will exercise at 40% MIP in the first week and 60% MIP in the subsequent five weeks. The patients will be instructed to inhale using the diaphragm muscle, trying to expand the rib cage to avoid using accessory muscles (Turqueto et al, 2021).

A nose clip will be used to ensure patients breathe exclusively through the training device. All patients will have their training sessions supervised by the same physical therapist and will be encouraged to maintain their usual activities during the protocol (Turqueto et al, 2021).

Control patients (CG), who will undergo muscle strengthening and aerobic training during pulmonary rehabilitation, will receive the same IMT intervention using POWERbreathe classic medic® (POWERbreathe International Limited, Southam, United Kingdom) soon after completion of the 6-week experimental protocol, if the study has satisfactory results.

STATISTICAL ANALYSIS Data normality will be tested through the Shapiro-Wilk test. To analyze the differences between groups, the t-test will be used for parametric data and the Wilcoxon test for non-parametric data. Bilateral tests will be performed using a significance level set at 5% (p < 0.05). Data will be analyzed using the SPSS 8.0 software and the results expressed as mean ± standard deviation or median and interquartile range.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes diagnosed with COVID-19 by RT-PCR who are not in the transmission window;
* Individuals between 30 and 70 years of age;
* A signed FICF.

Exclusion Criteria:

* Patients who had previously undergone IMT;
* Inability to perform the assessment tests;
* Orthopedic, visual, and neurological problems that would limit exercise treatment;
* Patients who are unable to undergo IMT because of discomfort with the use of the device;
* Respiratory diseases, severe heart and/or neuromuscular diseases that pre-exist COVID-19;
* Participants who do not have 90% attendance at rehabilitation sessions;
* Patients who required orotracheal intubation and use of mechanical ventilation support;
* Patients with body mass index (BMI) above 40.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
MIP assessment | 6 weeks
  This measurement, obtained by means of a digital manovacuometer (POWERbreathe K series KH2®, HaB International, Warwickshire, United Kingdom), reflects the pressure developed by the respiratory muscles plus the elastic recoil pressure of the respiratory system in the residual volume and is an index of global respiratory output rather than a direct measure of the contractile properties of the inspiratory muscles. This result will be used to monitor the influence of IMT on inspiratory muscle strength.
  The present proposal will predict MIP values through the equation of Neder et al., in which:
  For men: MIP (cmH2O) = 155,3 - (0,80 x age) For women: MIP (cmH2O) = 110,4 - (0,49 x age)

SECONDARY OUTCOMES:
S-Index assessment | 6 weeks
  The S-Index is a measure of the dynamic strength of the inspiratory muscles and is derived from the result of the peak inspiratory flow registered by the sensors of the device (POWERbreathe K series KH2®, HaB International, Warwickshire, United Kingdom) in each incursion, using a patented algorithm. Unlike the isometric measurement (MIP), in this assessment the individual will perform the inspiratory maneuver through a valve with free air passage. Inspiratory muscle strength is calculated across the entire range of inspired lung volume. The result of the strength index is classified based on the normal values predicted for the population studied. These values, which are recorded in cmH2O, are individually calculated by the software Breathelink® (POWERbreathe, Warwickshire, United Kingdom), using information from the patient's profile.
Assessment of inspiratory muscle endurance | 6 weeks
  Endurance - which is the ability to sustain a specific task over time - will be assessed using the electronic device POWERbreathe K series KH2®, HaB International, Warwickshire, United Kingdom) as a tool (POWERbreathe, 2019). The training load will be predetermined manually and introduced gradually over the first five breaths, as this is a constant load test, at 60% of the MIP value obtained from each patient. The patient will be instructed to breathe as long as possible until no breath can be fully completed, that is, until respiratory fatigue occurs. In the absence of respiratory fatigue, the maximum evaluation limit will be seven minutes, when the test is successfully completed. The results of resistance training will be recorded in the software and include the following parameters: Time (min), Peak Inspiratory Flow (l/s), Training Load (cmH2O), Average Power (Watts), Average Inspired Volume (l), and Energy (Joules).
1-MINUTE SIT-TO-STAND TEST | 6 weeks
  This test assesses the functional capacity of individuals with different types of diseases or dysfunctions. This standardized assessment is performed in an armless, 46-cm-high chair. The individual evaluated receives the verbal command to get up and sit down from the chair as many times as possible within a 1-minute interval. The main outcome of the test is how many times the individual sat and stood up; secondarily, vital and perceived exertion data are recorded before, during, and immediately after the test is performed.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Maurício Bona Gracelli, Vila Velha, Espírito Santo
  - Maurício Bona Gracelli, Vitória, Espírito Santo